CLINICAL TRIAL: NCT05445102
Title: Clinical and Radiographic Effect of Extracted Autogenous Demineralized Dentin as a Bone Graft Substitute in Management of Periodontal Intrabony Defects: A Case Series
Brief Title: Effect of Autogenous Demineralized Dentin as a Bone Graft Substitute in Management of Periodontal Intrabony Defects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Mohamed Shehata Abde Elmonaem, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11422
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Intrabony Defect
MeSH Terms: interventions — Bone Substitutes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- autogenous demineralized dentin graft as bone substitute in treatment of intrabony defect (Experimental)
  Interventions: Procedure: autogenous demineralized dentin graft as bone substitute in treatment of intrabony defect

INTERVENTIONS:
Procedure: autogenous demineralized dentin graft as bone substitute in treatment of intrabony defect — after extraction of tooth it will be grinded using hand bone mill and demineralized and placed in intrabony defect

SUMMARY:
one of the ultimate goals in periodontology is to achieve periodontal regeneration and change the prognosis of questionable or hopeless teeth to maintainable.Bone substitutes have been actively used to reconstruct bony defects. Four categories of bone graft materials exist: Autograft, Allograft, Alloplast, and Xenograft.many researchers paid attention to human tooth as one of the intraoral donor sites due to the chemical and structural similarity between dentin and alveolar bone since both demonstrate low crystalline hydroxyl appetite (HA) with comparable calcium-to-phosphorus ratio.

Extracted tooth will be cleaned from periodontal ligaments, cementum, soft tissue attachment, caries, or restorations (if present), using a high-speed fine finishing stone and saline irrigation. The pulp chamber will be cleaned with sterile endodontic files. Subsequently, teeth will be grounded, using hand bone mill .

ADDG particles prepared by demineralization of tooth particles in 0.6N hydrochloric acid for 30 min to achieve demineralized then washed twice in saline and dried with sterile gauze. The intrabony defect will be debrided using hand and ultrasonic devices and then ADDG particles will fill the defect. Vertical or horizontal mattress sutures and additional interrupted single sutures will be performed to obtain primary closure of the interdental space. The selection of the suturing technique will be based upon the dimension of the interdental space and the thickness and height of the interdental tissues using 5-0 proline suture then follow up period at 3 months and 6 months measuring CAL which is primary outcome and radiographic bone fill , probing depth and recession which are secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

Motivated patient 18 years of age or order.

* Patient consulting in the outpatient clinic.
* Patient ready to perform oral hygiene instructions.
* Provide informed consent.
* Accepts the 6 months follow-up period.

Teeth related criteria:

* Tooth with one or two walled intra-bony defect, probing depth ≥ 5mm with intra osseous defect ≥ 3mm.
* Mature permanent tooth.
* Unrestorable tooth or fractured tooth beyond restoration, impacted third molar or Supernumerary tooth to be extracted and used as whole tooth graft inside the defect

Exclusion Criteria:

* Patient-related criteria:

  * Medically compromised patients.
  * Pregnant women.
  * Uncooperative patients.
  * Smokers.
  * Systemic diseases that may compromise healing or bone metabolism (e.g diabetes, hyperthyroidism)

Teeth related criteria:

* Teeth with supra-bony defects.
* Teeth with grade III mobility.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-05-22 (Actual); Primary Completion 2023-05-22 (Estimated); Study Completion 2023-09-22 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level gain | change from baseline at 3 month and change from baseline at 6 month
  measured by william's periodontal probe

SECONDARY OUTCOMES:
Probing depth | change from baseline at 3 month and at 6 month
  measured by William's periodontal probe
Radiographic bone fill | change from baseline at 3 month and at 6 month
  periapical radiograph using Digora system
Recession | change from baseline at 3 month and at 6 month
  measured by William's periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: weam Elbattway, doctor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt